CLINICAL TRIAL: NCT03810118
Title: Rate of Fluid Challenge Administration and Fluid Responsiveness: an Open-label, Multicentric, Randomized Clinical Trial.
Brief Title: Fluid Challenge Infusion and Response
Acronym: REFILL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Antonio Messina, ICU senior consultant, Humanitas Clinical and Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REFILL
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Neurosurgery; Cardiovascular System; Anesthesia, General

STUDY DESIGN:
Intervention Model Description: A single group of patient will receive 4 ml/kg fluid challenge in either 10 or 20 minutes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All the enrolled patients will receive the same mini-fluid challenge test of 100ml and then will complete the 4 ml/kg fluid challenge in either 10 or 20 minutes
  Interventions: Diagnostic Test: fluid challenge

INTERVENTIONS:
Diagnostic Test: fluid challenge — 4 ml/kg fluid challenge infused over in either 10 or 20 minutes

SUMMARY:
It is unclear if the rate of administration of the fluid challenge could affect the rate of fluid responsiveness.

The role of this small-dose (the so called mini-FC) has been recently tested to assess if the infusion of a small amount of fluids (100 ml in 1 minute) could predict the final effect of the residual aliquot (i.e., 250 ml of FC test subdivided as follows: 100 ml in 1 minute and 150 ml in 9 minutes). Both the sudden increase in the stroke volume and the reduction of PPV and SVV after a bolus of 100 ml of crystalloids administered in 1 minute showed high sensitivity and specificity in predicting the final outcome of the FC.

The primary aim of the present study is assess whether the does the rate of infusion of fluid challenge affect fluid responsiveness in neurosurgical supine patients.

The secondary aim is to assess the reliability of the changes in SV, PPV and SVV after a mini-FC test in predicting the final fluid responsiveness.

DETAILED DESCRIPTION:
Dedicated algorithms and protocols of anaesthetic care regarding fluid therapy are key factors to prevent perioperative hypovolaemia and/or hypervolemia, which are known to increase morbidity and length of hospital stay.

Fluid therapy is commonly used in critically ill and surgical patients to restore hemodynamics. The aim of volume expansion is to increase cardiac index and oxygen delivery and to improve tissue oxygenation. However, this occurs only in a situation of preload dependency (i.e. when the ventricle operates on the steep part of the Frank-Starling's curve). Moreover, giving fluids to a non-volume-responsive patient (preload independency) can result in detrimental pulmonary and interstitial oedema. Fluid responsiveness (i.e., increase in stroke volume, SV, after fluid challenge, FC, administration) can be detected in 35-50% of both critically ill and surgical patients. The FC consists in assessing the hemodynamic effects of giving a small amount of fluid in a short period of time. The FC allows restoring fluid depletion when indicated, while minimizing the risk of overloading, which makes it the gold standard for assessing fluid depletion in patients undergoing surgery.

Then, FC administration should be based on predictors of fluid responsiveness. Static indexes, such as the central venous pressure, do not seem appropriate, whereas dynamic indexes, such as pulse pressure variation (PPV) and stroke volume variation (SVV), reliably predict the effect of FC administration during controlled mechanical ventilation only in case of a tidal volume (VT) of at least 8 mL/kg, which unfortunately are rarely found in both critically ill and surgical patients.

To overcome this VT-related limitation of PPV and SVV, the prediction of fluid responsiveness can be also achieved by applying functional hemodynamic tests aiming at increasing venous return and enhancing right ventricle preload dependence.

For example, when a FC is performed using a rapid infusion rate and a relatively "small" dose, its effect is sufficient to test whether the patient is on the ascending part of the cardiac function curve, hence showing an increase in cardiac output (CO).

The role of this small-dose (the so called mini-FC) has been recently tested to assess if the infusion of a small amount of fluids (100 ml in 1 minute) could predict the final effect of the residual aliquot (i.e., 250 ml of FC test subdivided as follows: 100 ml in 1 minute and 150 ml in 9 minutes). Both the sudden increase in the stroke volume and the reduction of PPV and SVV after a bolus of 100 ml of crystalloids administered in 1 minute showed high sensitivity and specificity in predicting the final outcome of the FC. However, the mini-FC has been tested, insofar, only in small-sized studies, needing further investigations to be confirmed.

Moreover, the response to the FC is transitory, and as such also its clinical effect. The study of Aya et al. pointed out that the effect of the FC is dissipated in about 10 minutes in both responders and non-responders and that a dose of 4 ml/kg of crystalloids is the lowest one to evocate a significant hemodynamic effect. It remains unclear, however, what the best approach to FC administration should be and, in fact, wide variability exists at this regard among studies performed both in the perioperative setting and in the intensive care unit (ICU). In fact, the rate of fluid administration is not fixed. A recent systematic review showed a significant heterogeneity. In a subgroup of 35 studies three (8.6%) reported an infusion rate of 1 ml/kg/min. In another group of 32 studies, the FC was administered in 30 minutes in 7 (21.8%) studies, in 20 minutes in 2 (6.2%) studies, in 13 minutes in 1 (3.1%) study, in 10 minutes in 15 studies (46.8%), in 5 minutes in 4 (12.5%) studies, in 3 minutes in 1 (3.1%) study, and in 2 minutes in 2 (6.2%) studies. The median (IQR) time of infusion was 10 (5-20) minutes.

After the indication of Aya et al., 4 ml/kg of crystalloids is the standard dose for the FC in our center. However, it is unclear if the rate of administration could affect the rate of fluid responsiveness. We, therefore, will perform a study to address this issue in a sample of neurosurgical patients.

The primary aim of the present study is assess whether the does the rate of infusion of fluid challenge affect fluid responsiveness in neurosurgical patients.

The secondary aim is to assess the reliability of the changes in SV, PPV and SVV after a mini-FC test in predicting the final fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged ≥ 18 years;
2. Scheduled for elective supine neurosurgery and requiring invasive arterial monitoring;
3. Glasgow coma scale 15 at recruitment

Exclusion Criteria:

1. Any recurrent cardiac arrhythmias;
2. Reduced left (ejection fraction <30%) or right (systolic peak velocity of tricuspid annular motion <0.17 m/s) ventricular systolic function;
3. Intra-operative use of vasopressors or inotropes before FC administration or between the first and the second bolus of fluids.
4. Chronic use beta-blocking agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Percentage of fluid responders | 10 or 20 minutes from the start
  Percentage of patients showing an increase in the stroke volume above the predefined threshold of fluid responsiveness after the infusion of the fluid challenge (>10%).
Pharmacodynamic effect of the FC | 10 or 20 minutes from the start
  AUC
Pharmacodynamic effect of the FC | 10 or 20 minutes from the start
  dmax
Pharmacodynamic effect of the FC | 10 or 20 minutes from the start
  Tmax
Pharmacodynamic effect of the FC | 10 or 20 minutes from the start
  d1
Pharmacodynamic effect of the FC | 10 or 20 minutes from the start
  d5

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mahjoub Y, Lejeune V, Muller L, Perbet S, Zieleskiewicz L, Bart F, Veber B, Paugam-Burtz C, Jaber S, Ayham A, Zogheib E, Lasocki S, Vieillard-Baron A, Quintard H, Joannes-Boyau O, Plantefeve G, Montravers P, Duperret S, Lakhdari M, Ammenouche N, Lorne E, Slama M, Dupont H. Evaluation of pulse pressure variation validity criteria in critically ill patients: a prospective observational multicentre point-prevalence study. Br J Anaesth. 2014 Apr;112(4):681-5. doi: 10.1093/bja/aet442. Epub 2013 Dec 29. PMID 24374504
- [Result] Biais M, de Courson H, Lanchon R, Pereira B, Bardonneau G, Griton M, Sesay M, Nouette-Gaulain K. Mini-fluid Challenge of 100 ml of Crystalloid Predicts Fluid Responsiveness in the Operating Room. Anesthesiology. 2017 Sep;127(3):450-456. doi: 10.1097/ALN.0000000000001753. PMID 28640019
- [Result] Muller L, Toumi M, Bousquet PJ, Riu-Poulenc B, Louart G, Candela D, Zoric L, Suehs C, de La Coussaye JE, Molinari N, Lefrant JY; AzuRea Group. An increase in aortic blood flow after an infusion of 100 ml colloid over 1 minute can predict fluid responsiveness: the mini-fluid challenge study. Anesthesiology. 2011 Sep;115(3):541-7. doi: 10.1097/ALN.0b013e318229a500. PMID 21792056
- [Result] Aya HD, Ster IC, Fletcher N, Grounds RM, Rhodes A, Cecconi M. Pharmacodynamic Analysis of a Fluid Challenge. Crit Care Med. 2016 May;44(5):880-91. doi: 10.1097/CCM.0000000000001517. PMID 26683506